CLINICAL TRIAL: NCT02703103
Title: Use of a New Mechanical Chest Compression Machine LifeLine ARM for Cardiopulmonary Resuscitation by Paramedics: a Randomized, Crossover, Manikin Trial
Brief Title: Chest Compression During Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Łukasz Szarpak, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02.008.1MR
Record Dates: First submitted 2016-02-16; First posted 2016-03-09 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: cardiopulmonary resuscitation; chest compression; adult; simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard cardiopulmonary resuscitation (Experimental): standard CPR (30:2) according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation.
  Interventions: Other: Manual chest compressions; Device: ARM chest compressions
- asynchronous cardiopulmonary resuscitation (Experimental): asynchronuos CPR according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation.
  Interventions: Other: Manual chest compressions; Device: ARM chest compressions

INTERVENTIONS:
Other: Manual chest compressions — 2 min of Chest compressions without mechanical chest compression system
Device: ARM chest compressions — 2 min of Chest compressions with mechanical chest compression system LifeLine ARM

SUMMARY:
The aim of the study was to evaluate the new mechanical chest compression machine LifeLine ARM in healthcare professionals in simulated model of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* maximum 1 year of work experience in medicine
* minimum 10 clinical resuscitations
* paramedics

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
chest compressions effectiveness | 1 day
  the percentage of correct chest compressions relative to the total number of chest compressions

SECONDARY OUTCOMES:
Depth | 1 day
  correct depth according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
Pressure point | 1 day
  correct pressure point according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
Complete pressure release | 1 day
  Complete pressure release measure by manikin software
Rate of chest compressions | 1 day
  correct chest compressions rate according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
hands-off time | 1 day
  defined as the sum of all periods during which no hand was placed on the chest minus time used for ventilation.
tidal volume | 1 day
  volume of air delivered in a single rescue breath in milliliters
ventilation rate | 1 day
  respiratory rate per minute
minute-volume | 1 day
  minute volume ventilation
number of gastric inflations | 1 day
  number of gastric inflations

CONTACTS AND LOCATIONS:
Locations (1):
- Łukasz Szarpak, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Truszewski Z, Szarpak L, Kurowski A, Evrin T, Zasko P, Bogdanski L, Czyzewski L. Randomized trial of the chest compressions effectiveness comparing 3 feedback CPR devices and standard basic life support by nurses. Am J Emerg Med. 2016 Mar;34(3):381-5. doi: 10.1016/j.ajem.2015.11.003. Epub 2015 Nov 4. PMID 26612703
- [Background] Kurowski A, Czyzewski L, Bogdanski L, Zasko P, Karczewska K, Szarpak L. Quality of chest compression with CardioPump CPR compared to single rescuer standard BLS. Am J Emerg Med. 2015 Jan;33(1):114-5. doi: 10.1016/j.ajem.2014.10.027. Epub 2014 Oct 20. No abstract available. PMID 25455057